CLINICAL TRIAL: NCT03001778
Title: Smart Television and Exercise Promotion for Independent Living Facilities
Acronym: STEP4Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21AG046670 (NIH); 5R21AG046670 (NIH); 0283 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Aging; Physical Activity
Keywords: Physical Activity; Older Adults; Independent Living Facilities; Multimedia technology
MeSH Terms: conditions — Motor Activity | interventions — User-Centered Design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usability Testing (Experimental): Prototype testing
  Interventions: Other: Usability Testing

INTERVENTIONS:
Other: Usability Testing — Usability testing of "ready made" workouts in a group format.

SUMMARY:
Physical activity (PA) has physical, emotional, and cognitive benefits for seniors (e.g., increased strength and balance, reduced frailty, fewer falls, improved brain function, lower mortality risk), yet many seniors have limited access to exercise options due to numerous barriers (e.g., transportation concerns, financial costs, fear of injury/falling). This project will overcome common exercise barriers by creating an interactive web-enabled TV program (i.e., Smart TV), adapted from research-based PA protocols, to be implemented in an Independent Living Facility (ILF) setting. A web-based prototype will be developed, and ILF residents and administrators will be able to create, use, and evaluate a customizable exercise program tailored to the individual's preferred type of exercise, intensity, and duration.

DETAILED DESCRIPTION:
Older Adults (OAs), aged 65 years and older, are the fastest growing segment of the U.S. population. As life expectancy increases, maintaining physical independence has become a public health priority. It is well recognized that regular physical activity (PA) can be done safely by seniors, and has multiple physical, emotional, and cognitive benefits. Yet, they remain the least physically active of any age group. This suggests that the translational reach of efficacious PA protocols to the real-world remains limited, and a need for research which is scalable to the individual in more naturalistic settings exists. An emerging trend for seniors is to choose Independent Living Facilities (ILFs) as their home. ILFs offer a variety of social, cultural, and fitness services. Access to up-to-date technologies (e.g., wireless Internet), web-based education, and wellness programs are a priority for ILF residents, thus opportunities for using technology for health promotion with OAs exists. ILFs provide a unique opportunity for PA promotion, because 1) more seniors are choosing ILFs for aging-in-place, 2) PA is of interest to ILF residents, 3) ILFs should continue to increase their wellness offerings, and 4) ILFs should be interested in incorporating PA programs into wellness offerings. Research is needed to translate efficacious PA protocols for seniors into formats that are scalable to OAs in real-world settings. The goal is to extrapolate knowledge gained from efficacy research to improve the utilization and sustainability of evidence-based methods by producing programs that are agreeable, user-friendly, and optimal at both the individual and organizational level. Smart Television and Exercise Promotion for Independent Living Facilities (STEP for LIFE) will establish the feasibility for translating an evidence-based PA program using an interactive web-enabled, streaming-video technology (i.e., Smart TV) for ILF residents. This program offers 1) an innovative and potentially effective medium to reach seniors, 2) the ability to select and sequence together a session that is personalized to fitness level, type of exercise, and duration, and 3) organizations the ability to provide desired wellness options which meet both resident and organizational needs. The purpose of this study is to provide the initial research for translating efficacious research-based PA protocols for seniors into a scalable format usable in a real-world ILF setting, and to gain knowledge at individual and organizational levels to improve implementation and sustainability of this evidence-based approach. Specific Aims include extensive formative research on the use, interest, and effectiveness of interactive multimedia approaches for promoting PA, and its integration into senior living settings. A working prototype will be developed and tested for usability with ILF residents and administrators, and seniors not residing in ILFs. Outcomes will establish the feasibility of producing and testing STEP for LIFE in a large-scale randomized trial. A larger trial can inform 1) future translation of PA promotion to other OA residential settings (e.g., assisted living, memory care, rural settings), and 2) sustainable implementation strategies for other evidence-based health promotion protocols for seniors.

ELIGIBILITY:
Independent Living Facility (ILF) Resident Inclusion Criteria:

* 55 years of age or older
* live in an ILF
* able tor read and speak English
* able to consent to participate
* exercise 60 min or more a week (self-reported)

ILF Resident Exclusion Criteria:

* under 55 years of age
* not live in an ILF
* unable to read and speak English
* unable to consent to participate
* exercise less than 60 minutes (self-reported)

Non-ILF Resident Inclusion Criteria:

* 55 years of age or older
* not live in an ILF
* able to read and speak English
* able to consent to participate
* exercise 60 min or more a week (self-reported)

Non-ILF Resident Exclusion Criteria:

* under 55 years of age
* live in an ILF
* unable to read and speak English
* unable to consent to participate
* exercise less than 60 minutes (self-reported)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PhD', Principal Investigator — Klein Buendel, Inc.
Locations (1):
- Klein Buendel, Inc., Golden, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan DC, Tsou HH, Yang RS, Tsauo JY, Chen CY, Hsiung CA, Kuo KN. A pilot randomized controlled trial to improve geriatric frailty. BMC Geriatr. 2012 Sep 25;12:58. doi: 10.1186/1471-2318-12-58. PMID 23009149
- [Background] Xue QL, Bandeen-Roche K, Mielenz TJ, Seplaki CL, Szanton SL, Thorpe RJ, Kalyani RR, Chaves PH, Dam TT, Ornstein K, RoyChoudhury A, Varadhan R, Yao W, Fried LP. Patterns of 12-year change in physical activity levels in community-dwelling older women: can modest levels of physical activity help older women live longer? Am J Epidemiol. 2012 Sep 15;176(6):534-43. doi: 10.1093/aje/kws125. Epub 2012 Aug 30. PMID 22935515
- [Background] Langlois F, Vu TT, Chasse K, Dupuis G, Kergoat MJ, Bherer L. Benefits of physical exercise training on cognition and quality of life in frail older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):400-4. doi: 10.1093/geronb/gbs069. Epub 2012 Aug 28. PMID 22929394
- [Background] Kamegaya T; Long-Term-Care Prevention Team of Maebashi City; Maki Y, Yamagami T, Yamaguchi T, Murai T, Yamaguchi H. Pleasant physical exercise program for prevention of cognitive decline in community-dwelling elderly with subjective memory complaints. Geriatr Gerontol Int. 2012 Oct;12(4):673-9. doi: 10.1111/j.1447-0594.2012.00840.x. Epub 2012 Apr 2. PMID 22469534
- [Background] Uemura K, Doi T, Shimada H, Makizako H, Yoshida D, Tsutsumimoto K, Anan Y, Suzuki T. Effects of exercise intervention on vascular risk factors in older adults with mild cognitive impairment: a randomized controlled trial. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):445-55. doi: 10.1159/000343486. Epub 2012 Oct 25. PMID 23189083
- [Background] Concannon LG, Grierson MJ, Harrast MA. Exercise in the older adult: from the sedentary elderly to the masters athlete. PM R. 2012 Nov;4(11):833-9. doi: 10.1016/j.pmrj.2012.08.007. PMID 23174546
- [Background] Rydwik E, Welmer AK, Kareholt I, Angleman S, Fratiglioni L, Wang HX. Adherence to physical exercise recommendations in people over 65--the SNAC-Kungsholmen study. Eur J Public Health. 2013 Oct;23(5):799-804. doi: 10.1093/eurpub/cks150. Epub 2012 Oct 31. PMID 23115329
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Background] Faber MJ, Bosscher RJ, Chin A Paw MJ, van Wieringen PC. Effects of exercise programs on falls and mobility in frail and pre-frail older adults: A multicenter randomized controlled trial. Arch Phys Med Rehabil. 2006 Jul;87(7):885-96. doi: 10.1016/j.apmr.2006.04.005. PMID 16813773
- [Background] Li F, Harmer P, Fisher KJ, McAuley E, Chaumeton N, Eckstrom E, Wilson NL. Tai Chi and fall reductions in older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2005 Feb;60(2):187-94. doi: 10.1093/gerona/60.2.187. PMID 15814861
- [Background] Spirduso WW, Cronin DL. Exercise dose-response effects on quality of life and independent living in older adults. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S598-608; discussion S609-10. doi: 10.1097/00005768-200106001-00028. PMID 11427784
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Mather AS, Rodriguez C, Guthrie MF, McHarg AM, Reid IC, McMurdo ME. Effects of exercise on depressive symptoms in older adults with poorly responsive depressive disorder: randomised controlled trial. Br J Psychiatry. 2002 May;180:411-5. doi: 10.1192/bjp.180.5.411. PMID 11983637
- [Background] Sze PC, Cheung WH, Lam PS, Lo HS, Leung KS, Chan T. The efficacy of a multidisciplinary falls prevention clinic with an extended step-down community program. Arch Phys Med Rehabil. 2008 Jul;89(7):1329-34. doi: 10.1016/j.apmr.2007.11.044. PMID 18586135
- [Background] Stevens JA, Sogolow ED. Preventing Falls: What Works: A CDC Compendium of Effective Community-Based Interventions From Around the World. National Center for Injury Prevention and Control; 2008.
- [Background] Najafi B, Armstrong DG, Mohler J. Novel wearable technology for assessing spontaneous daily physical activity and risk of falling in older adults with diabetes. J Diabetes Sci Technol. 2013 Sep 1;7(5):1147-60. doi: 10.1177/193229681300700507. PMID 24124940
- [Background] Gschwind YJ, Kressig RW, Lacroix A, Muehlbauer T, Pfenninger B, Granacher U. A best practice fall prevention exercise program to improve balance, strength / power, and psychosocial health in older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2013 Oct 9;13:105. doi: 10.1186/1471-2318-13-105. PMID 24106864
- [Background] Lee H, Lee JA, Brar JS, Rush EB, Jolley CJ. Physical activity and depressive symptoms in older adults. Geriatr Nurs. 2014 Jan-Feb;35(1):37-41. doi: 10.1016/j.gerinurse.2013.09.005. Epub 2013 Oct 18. PMID 24144579
- [Background] National Prevention Council, Health Promotion Council, Public Health Council. Active Living. The National Prevention Strategy. http://www.surgeongeneral.gov/initiatives/prevention/strategy/report.html. June 16, 2011.
- [Background] Schillinger D. An introduction to effectiveness, dissemination and implementation research. In: Fleisher P, Goldstein E, editors. San Francisco: Clinical Translational Science Institute Community Engagement Program, University of California San Francisco; 2010.
- [Background] Koh HK. A 2020 vision for healthy people. N Engl J Med. 2010 May 6;362(18):1653-6. doi: 10.1056/NEJMp1001601. No abstract available. PMID 20445177
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] U.S.Department of Health and Human Services. 2008 physical activity guidelines for Americans. Be active, healthy, and happy. Publication No.U0036 http://www.health.gov/paguidelines/. 2008.
- [Background] The Society of Certified Senior Advisors. State of the senior housing industry. The Society of Certified Senior Advisors Web site. http://www.csa.us/docs/StateoftheSeniorHousingIndustryReport.pdf. 2011.
- [Background] Brecht S, Fein S, Hollinger-Smith L. Preparing for the future: trends in continuing care retirement communities. Seniors Housing & Care Journal. 2009;17(1):75-90.
- [Background] Mather Lifeways Institute on Aging. Trend survey reveals future of senior living communities. http://matherlifeways.com/archives/1373. May 19, 2009.

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Residents: Community prototype testing
  Usability Testing: Usability testing of "ready made" workouts.
- ILF Resident Usability Testing: ILF Prototype testing
  Usability Testing: Usability testing of "ready made" workouts.
Period: Overall Study
Arm/Group | Community Residents | ILF Resident Usability Testing
Started | 21 | 46
Completed | 21 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Community Usability Testing: Prototype testing
  Usability Testing: Usability testing of "ready made" workouts in a group format.
- ILF Usability Testing: Prototype testing
  Usability Testing: Usability testing of "ready made" workouts in as an individual.
- Total: Total of all reporting groups
Arm/Group | Community Usability Testing | ILF Usability Testing | Total
Number analyzed (Participants) | 21 | 46 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 33 | 41
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 45 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 46 | 67

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (SUS)
Description: Ten likert-type questions assessing user-friendliness of technology. Each question has five answer options that range from "Strongly Agree" to "Strongly Disagree". Scores range from 0-100. A score of 68 or above is considered above average. All scores averaged.
Time Frame: After 1 hour usability session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community Residents | ILF Resident Usability Testing
Number analyzed (Participants) | 21 | 46
units on a scale | 73.57 (22.12) | 74.70 (13.94)

ADVERSE EVENTS:
Time Frame: 1 year 6 months
Groups:
- Community Usability Testing; ILF Usability Testing: Prototype testing
  Usability Testing: Usability testing of "ready-made" workouts in a group format.
Arm/Group | Community Usability Testing | ILF Usability Testing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/46
Other Adverse Events (participants affected / at risk) | 0/21 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-08-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03001778/SAP_000.pdf
  • Study Protocol (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03001778/Prot_001.pdf